CLINICAL TRIAL: NCT04431791
Title: A Single-center，Observational，Ambispective Cohort Study of Regorafenib Versus Fruquintinib in Metastatic Colorectal Cancer Patients Who Have Progressed After at Least Second Lines of Chemotherapies
Brief Title: Real World Study of Regorafenib Versus Fruquintinib in Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, MD, Professor, Chief of Department of GI Oncology, Peking University Cancer Hospital, Peking University
Other Study IDs: Reg vs Fru
Record Dates: First submitted 2020-06-06; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Colorectal Cancer
Keywords: Targeted therapy; TTF; OS; PFS; AE
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib; HMPL-013

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Regorafenib
  Interventions: Drug: Regorafenib
- Fruquintinib
  Interventions: Drug: Fruquintinib

INTERVENTIONS:
Drug: Regorafenib — oral regorafenib
  Groups: Regorafenib
Drug: Fruquintinib — oral fruquintinib
  Groups: Fruquintinib

SUMMARY:
This is an observational, ambispective cohort study. The aim is to compare the efficacy and safety of regorafenib versus fruquintinib conducted in China. About 268 eligible metastatic colorectal cancer patients after second-line therapy will be assigned to receive either regorafenib or fruquintinib, based on decision of the gastrointestinal physician according the patients' condition.

ELIGIBILITY:
Inclusion Criteria:

1. signed and dated informed consent.
2. Diagnosis of histologically confirmed colorectal cancer, stage IV.
3. after second-line therapy.
4. gastrointestinal physician prescribed to receive regorafenib or fruquintinib according the patients' condition.

Exclusion Criteria:

1. received regorafenib or fruquintinib before third-line therapy.
2. the clinicopathological characteristics and previous therapy were unknown.
3. regorafenib or fruquintinib treatment is less than one cycle in the historical cohort.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with signing the informed consent, would be enrolled when their gastrointestinal physician prescribed to receive regorafenib or fruquintinib after second-line according the condition.
Sampling Method: Non-Probability Sample
Enrollment: 268 (Estimated)
Dates: Start 2020-05-25 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Time To Treatment Failure | every month, up to discontinuation of treatment for any reason.
  the time from first dose to discontinuation of treatment for any reason, including disease progression, treatment toxicity, and death.

SECONDARY OUTCOMES:
Overall survival | from enrollment of the first subject until the database cut-off approximately 6 months later.
  the time from first dose to the death for any cause.
Progression-free survival | from enrollment of the first subject until the database cut-off approximately 6 months later.
  the time from first dose to disease progression.
Incidence of adverse events（AEs） | from the first dose to discontinuation of treatment for any reason, including disease progression, treatment toxicity, and death.
  percentage of patients with AEs according to CTCAE 4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China